CLINICAL TRIAL: NCT06840275
Title: A Danish, Double-blind, Randomized Placebo-controlled Clinical Trial Evaluating Allogeneic Adipose Tissue Derived Mesenchymal Stromal Cell Therapy in Patients With Recently Diagnosed Non-ishemic Heart Failure With Reduced Ejection Fraction
Brief Title: ASCs in Recently Diagnosed Non-ischemic Heart Failure
Acronym: ARIISE
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cell to Cure ApS (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ARIISE; 2025-520837-22-00 (EU CTIS Number); U1111-1315-7011 (Other: WHO universal trial number)
Record Dates: First submitted 2025-02-03; First posted 2025-02-21 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Non-Ischemic Heart Failure; Reduced Ejection Fraction Heart Failure
Keywords: allogeneic adipose tissue derived mesenchymal stromal cell; non-ischemic heart failure; mesenchymal stromal cell
MeSH Terms: conditions — Heart Failure, Systolic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Allogeneic adipose tissue-derived mesenchymal stromal cells (C2C_ASC110) (Experimental): Intravenous infusion of allogeneic adipose tissue-derived mesenchymal stromal cells (C2C_ASC110) 1 month apart.
  Interventions: Drug: Allogeneic adipose tissue-derived mesenchymal stem cells
- CryoStor® CS10 (Placebo Comparator): Intravenous infusion of CryoStor® CS10 1 month apart.
  Interventions: Other: Cryostor CS10

INTERVENTIONS:
Drug: Allogeneic adipose tissue-derived mesenchymal stem cells — Two intravenous infusions of C2C_ASC110 1 month apart. The C2C_ASC110 product contains 110 million cells.
  Other Names: C2C_ASC110
  Arms: Allogeneic adipose tissue-derived mesenchymal stromal cells (C2C_ASC110)
Other: Cryostor CS10 — Two intravenous infusions of CryoStor CS10 1 month apart.
  Arms: CryoStor® CS10

SUMMARY:
The goal of this clinical trial is to investigate the efficacy and safety of intravenous infusions of allogeneic adipose tissue-derived mesechymal stromal cells in patients with recently diagnosed non-ischemic heart failure in restoring cardiac function compared to placebo. The primary outcome of this trial is the change in left ventricular ejection fraction 6 month after treatment compared to placebo. Participants will be given two treatments with one month apart of either allogeneic adipose tissue-derived mesechymal stromal cells or placebo.

DETAILED DESCRIPTION:
Non-ischemic heart failure (NIHF) is the leading reason for heart transplantation. The disease can be caused by several different factors, which include genetic disposition, inflammation, hypertension, alcohol consumption, and arrhythmia. Regardless of the aetiology, immune activation in myocardium leads to collagen deposition and decreases the function of heart. There are currently no treatment options, which reverse the inflammatory component in NIHF.

For the past decade, cell therapy has been tested as treatment option for ischemic and non-ischemic heart failure. Especially the mesenchymal stromal cell (MSC) has shown encouraging results for their potential to improve cardiac function in patients with non-ischemic heart failure along with its safety. The cardiac improvement may be related to the immunomodulation as MSC is known by its ability to modulate the immune system and has successfully been applied clinically as a novel active immunosuppressor.

We aim to conduct a clinical trial in which patients recently diagnosed with NIHF will be randomized to either treatment with two intravenous infusions of allogeneic MSCs obtained from adipose tissue (C2C_ASC110) or placebo (Cryostor® CS10) 4 weeks apart. The objective is to evaluate the safety and effect of MSCs on cardiac function.

The long-term perspective is that the information gathered from this study can lead to a new treatment option for this specific group of patients, who currently have no further treatment options and a poor prognosis.

ELIGIBILITY:
Inclusion Criteria:

* Patients above 18 years of age
* Written informed consent
* Anticipated to be able to participate during the entire study period
* Diagnosed with non-ischemic heart failure with initial LVEF ≤ 40% and then up-titrated to maximal tolerable heart failure medication within the last 12 months
* Symptomatic heart failure (NYHA II-III)
* LVEF ≤ 45 % documented by echocardiography, CT or MRI performed after up-titration of heart failure medication (documentation of reduced LVEF at least after 1 and 3 months if implantation of a device either an Implantable Cardioverter Defibrillator (ICD) or Cardiac Resynchronisation Therapy (CRT), respectively)
* Plasma Pro-BNP > 300 pg/ml (> 35 pmol/L) in patients with sinus rhythm and plasma Pro-BNP > 422 pg/ml (> 49 pmol/L) in patients with atrial fibrillation.

Exclusion Criteria:

* NYHA I or IV heart failure
* Documented ischemic heart failure
* On-going alcohol abuse
* Implantation of CRT within 3 months or ICD within 1 month
* Acute coronary syndrome with elevation of CKMB (Creatine Phosphatase-Myocardial Band) or troponins, stroke or transitory cerebral ischemia within six weeks of inclusion
* Expected to undergo screening for heart transplantation during the study time
* Listed for heart transplantation
* Other cardiac revascularization treatments to be performed
* Moderate to severe aortic stenosis (valve area < 1.1 cm2) or clinically significant mitral valve disease
* Diminished functional capacity for other reasons such as: chronic obstructive pulmonary disease (COPD) with forced expiratory volume (FEV) < 1 L/min or body mass index > 35kg/m2
* Clinically significant anaemia (haemoglobin < 6 mmol/L), leukopenia (leucocytes < 2 109/L), leucocytosis (leucocytes >14 109/L) or thrombocytopenia (thrombocytes < 50 109/L)
* History with malignant disease within five years of inclusion or current suspected malignancy - except treated skin cancer other than melanoma
* Patients with known hypersensitivity to DMSO and Dextran-40.
* Pregnant women
* Other experimental treatment within four weeks from baseline tests
* Participation in another interventional trial

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2028-09-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
Change in left ventricular ejection fraction (I) | From enrollment to 6 months after the last infusion of C2C_ASC110 and placebo.
  Change in left ventricular ejection fraction 6 months after last C2C_ASC110 infusion compared to the placebo group.

SECONDARY OUTCOMES:
Changes in left ventricular end systolic volume | From enrollment to 7 months and to 12 months.
  Changes in left ventricular end systolic volume
Change in left ventricular ejection fraction (II) | From enrollment to 7 months and to 12 months.
  Change in left ventricular ejection fraction.
Changes in left ventricular end diastolic volume | From enrollment to 7 months and to 12 months.
  Changes in left ventricular end diastolic volume.
Change in NYHA classification | From enrollment to 12 months.
  Change in New York Heart Association (NYHA) classification. A scale from 1 to 4 describing the extent of heart failure by patient-reported symptoms, with class 1 denoting no symptoms and no limitations in ordinary physical activity and class 4 denoting symptoms and severe limitations in ordinary physical activity.
Change in KCCQ questionnaire score | From enrollment to 12 months.
  Change in Kansas City Cardiomyopathy (KCCQ) questionnaire score. A scale from 0 to 100 describing health status in patients with heart failure, with 0 denoting the worst possible health status and 100 denotes the best possible health status.
Change in EQ5D5L questionnaire score | From enrollment to 12 months.
  Change in European Quality of Life - 5 Dimensions (EQ5D5L) questionnaire score. A scale from 0 to 100 describing health related quality of life, with 0 denoting the worst possible quality of life and 100 denoting the best possible quality of life.
Change in 6 minutes walking test | From enrollment to 12 months.
  Change in 6 minutes walking test.
Change in Pro-BNP | From enrollment to 12 months.
  Change in Pro-BNP.
Incidence and severity of adverse reactions | From the first infusion of C2C_ASC110 and placebo to 12 months.
  Incidence and severity of serious adverse reactions and suspected unexpected serious adverse reactions.

CONTACTS AND LOCATIONS:
Overall Officials: Abbas A Qayyum, MD MSc PhD, Principal Investigator — Cardiology Stem Cell Centre, Department of Cardiology, The Heart Centre, Rigshospitalet, Copenhagen
Locations (1):
- Cardiology Stem Cell Centre, Department of Cardiology, The Heart Centre, Rigshospitalet, University of Copenhagen, Denmark, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No